CLINICAL TRIAL: NCT05608109
Title: Project Smash (Social Media Alcohol Session for Health)
Brief Title: A Social Media Personalized Normative Feedback Intervention for Heavy Drinking College Students
Acronym: SMASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/05/12; R00AA025394 (NIH)
Record Dates: First submitted 2022-10-24; First posted 2022-11-08 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-11

CONDITIONS: Alcohol Consumption
Keywords: social media
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Alcohol personalized normative feedback (APNF) (Experimental): Participants will receive feedback about their consumption, what they think the average student at their university drinks, and actual drinking statistics at their university.
  Participants in this condition will participate in a baseline survey and afterwards will receive the feedback intervention. They will then complete follow-up surveys at 3-months and 6-months.
  Interventions: Behavioral: Alcohol personalized normative feedback (APNF)
- Social media personalized normative feedback (SMPNF) (Experimental): Participants will receive feedback about their consumption and alcohol related consumption posts, what they think the average student at their university drinks, and actual drinking statistics at their university.
  Participants in this condition will participate in a baseline survey and afterwards will receive the feedback intervention. They will then complete follow-up surveys at 3-months and 6-months.
  Interventions: Behavioral: Social media personalized normative feedback (SMPNF)
- Alcohol and social media personalized normative feedback (APNF + SMPNF) (Experimental): Participants will go through the alcohol personalized normative feedback process and the social media personalized normative feedback.
  Participants in this condition will participate in a baseline survey and afterwards will receive the feedback intervention. They will then complete follow-up surveys at 3-months and 6-months.
  Interventions: Behavioral: Alcohol personalized normative feedback (APNF); Behavioral: Social media personalized normative feedback (SMPNF)
- Attention control (No Intervention): Participants will receive feedback about their consumption of desserts, what they think their peers consume, and actual dessert consumption statistics are for individuals in their age group in the United States.
  Participants in this condition will participate in a baseline survey/feedback intervention. They will then complete follow-up surveys and feedback interventions at 3-months and 6-months.

INTERVENTIONS:
Behavioral: Alcohol personalized normative feedback (APNF) — Participants will receive individualized feedback based upon their survey responses. Feedback regarding participant's drinking compared to other same-university students will include: (a) drinking days per week, (b) average drinks per occasion, (c) drinks per week, and (d) drinking percentile rank.
  Arms: Alcohol and social media personalized normative feedback (APNF + SMPNF); Alcohol personalized normative feedback (APNF)
Behavioral: Social media personalized normative feedback (SMPNF) — Participants will receive individualized feedback based upon their survey responses. Feedback regarding participant's alcohol related content posts on social media and drinking compared to other same-university students will include: (a) alcohol related posting days per week, (b) average alcohol related posting per week, (c) posting percentile rank, (d) drinking days per week, (e) average drinks per week, and (f) drinking percentile rank.
  Arms: Alcohol and social media personalized normative feedback (APNF + SMPNF); Social media personalized normative feedback (SMPNF)

SUMMARY:
This study seeks to evaluate the unique and synergistic efficacy of social media-specific personalized normative feedback targeting the reduction of alcohol use among heavy-drinking college students who post alcohol-related content on social media.

Hypothesis: Alcohol personalized normative feedback, social media-specific personalized normative feedback, and the Alcohol personalized normative feedback+ social media-specific personalized normative feedback conditions will be more effective in reducing drinking than the attention control condition.

ELIGIBILITY:
Inclusion Criteria:

* College students recruited across three universities: Duquesne University, Miami University, and University of Houston (DU, MU, UH)
* Undergraduate college students 18 to 26 years old
* Meet heavy drinking (4+ drinks in one sitting for individuals assigned female at birth, 5+ drinks in one sitting for individuals assigned male at birth in the past month) and ARC (alcohol-related content) posting criteria (2+ ARC posts in the last 30 days for individuals assigned female at birth, 1+ for individuals assigned male at birth, on either Facebook, Instagram, Snapchat, Twitter, or TikTok)

Exclusion Criteria:

* Pregnant or of another protected population

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 401 (Actual)
Dates: Start 2022-01-09 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Brief Young Adult Alcohol Consequences Questionnaire (B-YAACQ) - change is being assessed | Baseline, 3 month follow-up, 6 month follow-up
  The B-YAACQ is a 24 item assessment which measures consequences in 8 domains over a given time frame. Subscales include: Social/Interpersonal, Academic/Occupational, Risky Behavior, Impaired Control, Poor Self-Care, Diminished Self-Perception, Blackout Drinking, and Physiological Dependence. Minimum value: 0; Maximum Value: 24; Higher scores indicate more alcohol-related problems.
Alcohol Use Disorder Identification Test (AUDIT) - change is being assessed | Baseline, 3 month follow-up, 6 month follow-up
  The AUDIT is a 10 item tool which assesses a participant's drinking habits and alcohol-related consequences. Minimum value: 0; Maximum Value: 40; Higher scores indicate worse outcomes. A score of 15 or more indicates the likelihood of alcohol dependence.
Rutgers Alcohol Problems Index (RAPI) -change is being assessed | Baseline, 3 month follow-up, 6 month follow-up
  The RAPI is a 25-item questionnaire that measures problem drinking. Items are rated on a 4-point Likert scale, ranging from none (0) to more than five times (4). Minimum value: 0; Maximum Value: 100; Higher scores indicate more alcohol-related problems.
Quantity/Frequency/Peak Index (QFI) -change is being assessed | Baseline, 3 month follow-up, 6 month follow-up
  The QFI consists of five items which assess participants' typical alcohol consumption patterns. Minimum value: 0; Maximum Value: 24; Higher scores indicate more alcohol use.
Daily Drinking Questionnaire (DDQ) -change is being assessed | Baseline, 3 month follow-up, 6 month follow-up
  The DDQ is a 9 item tool which assesses participants' drinking over the past 3 months. Participants report how much they drank on an average over the past 3 months by indicating the number of drinks they consumed on each day of the week. Minimum value: 0; Maximum Value: 175 (windsorized to 25 drinks per day); Higher scores indicate more alcohol use.
Drinking Norms Rating Form (DNRF) -change is being assessed | Baseline, 3 month follow-up, 6 month follow-up
  The DNRF is a 5 item questionnaire that assesses an individual's view on the drinking habits of other individuals attending the same university. It was adapted from the Daily Drinking Questionnaire to assess perceptions of drinking norms on campus. Minimum value: 0; Maximum Value: 175 (windsorized to 25 drinks per day); Higher scores indicate students perceive their peers to engage in more alcohol use.

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Ly N Steers, PhD, Principal Investigator — Duquesne University
Locations (3):
- United States (3):
  - Miami University, Oxford, Ohio
  - University of Houston, Houston, Pennsylvania
  - Duquesne University, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wallace JM Jr, Bachman JG, O'Malley PM, Schulenberg JE, Cooper SM, Johnston LD. Gender and ethnic differences in smoking, drinking and illicit drug use among American 8th, 10th and 12th grade students, 1976-2000. Addiction. 2003 Feb;98(2):225-34. doi: 10.1046/j.1360-0443.2003.00282.x. PMID 12534428
- [Background] Rinker DV, Diamond PM, Walters ST, Wyatt TM, DeJong W. Distinct Classes of Negative Alcohol-Related Consequences in a National Sample of Incoming First-Year College Students: A Latent Class Analysis. Alcohol Alcohol. 2016 Sep;51(5):602-8. doi: 10.1093/alcalc/agw036. Epub 2016 Jun 20. PMID 27325885
- [Background] Curtis BL, Lookatch SJ, Ramo DE, McKay JR, Feinn RS, Kranzler HR. Meta-Analysis of the Association of Alcohol-Related Social Media Use with Alcohol Consumption and Alcohol-Related Problems in Adolescents and Young Adults. Alcohol Clin Exp Res. 2018 Jun;42(6):978-986. doi: 10.1111/acer.13642. Epub 2018 May 22. PMID 29786874
- [Background] Collins RL, Parks GA, Marlatt GA. Social determinants of alcohol consumption: the effects of social interaction and model status on the self-administration of alcohol. J Consult Clin Psychol. 1985 Apr;53(2):189-200. doi: 10.1037//0022-006x.53.2.189. No abstract available. PMID 3998247
- [Background] Read JP, Kahler CW, Strong DR, Colder CR. Development and preliminary validation of the young adult alcohol consequences questionnaire. J Stud Alcohol. 2006 Jan;67(1):169-77. doi: 10.15288/jsa.2006.67.169. PMID 16536141
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Martens MP, Neighbors C, Dams-O'Connor K, Lee CM, Larimer ME. The factor structure of a dichotomously scored Rutgers Alcohol Problem Index. J Stud Alcohol Drugs. 2007 Jul;68(4):597-606. doi: 10.15288/jsad.2007.68.597. PMID 17568966
- [Background] Dimeff, L. A. (Ed.). (1999). Brief alcohol screening and intervention for college students (BASICS): A harm reduction approach. Guilford Press.
- [Background] Lindgren KP, Neighbors C, Teachman BA, Baldwin SA, Norris J, Kaysen D, Gasser ML, Wiers RW. Implicit alcohol associations, especially drinking identity, predict drinking over time. Health Psychol. 2016 Aug;35(8):908-918. doi: 10.1037/hea0000396. PMID 27505215
- [Background] Cooper ML. Motivations for alcohol use among adolescents: development and validation of a four-factor-model. Psychological Assessment. 1994; 6(2): 117-128.
- [Background] Przybylski, AK, Murayama, K, DeHaan, CR, Gladwell, V. Motivational, emotional, and behavioral correlates of fear of missing out. Computers in Human Behavior. 2013; 29: 1814-1848.
- [Background] Shensa A, Sidani JE, Escobar-Viera CG, Switzer GE, Primack BA, Choukas-Bradley S. Emotional support from social media and face-to-face relationships: Associations with depression risk among young adults. J Affect Disord. 2020 Jan 1;260:38-44. doi: 10.1016/j.jad.2019.08.092. Epub 2019 Aug 29. PMID 31493637
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Radloff, LS. The CES-D Scale: A self-report depression scale for research in the general population. Applied Psychological Measurement. 1977; 1(3): 385-401.
- [Background] Lang FR, John D, Ludtke O, Schupp J, Wagner GG. Short assessment of the Big Five: robust across survey methods except telephone interviewing. Behav Res Methods. 2011 Jun;43(2):548-67. doi: 10.3758/s13428-011-0066-z. PMID 21424189
- [Background] Hays RD, DiMatteo MR. A short-form measure of loneliness. J Pers Assess. 1987 Spring;51(1):69-81. doi: 10.1207/s15327752jpa5101_6. PMID 3572711
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Andreassen CS, Torsheim T, Brunborg GS, Pallesen S. Development of a Facebook Addiction Scale. Psychol Rep. 2012 Apr;110(2):501-17. doi: 10.2466/02.09.18.PR0.110.2.501-517. PMID 22662404
- [Background] Baer JS, Stacy A, Larimer M. Biases in the perception of drinking norms among college students. J Stud Alcohol. 1991 Nov;52(6):580-6. doi: 10.15288/jsa.1991.52.580. PMID 1758185
- [Background] Sobell LC, Sobell MB. 2012. Timeline Follow-Back. In: Litten R.Z., Allen J.P. (eds) Measuring Alcohol Consumption. Humana Press, Totowa, NJ. https://doi.org/10.1007/978-1-4612-0357-5_3
- [Background] Zimmerman GL, Olsen CG, Bosworth MF. A 'stages of change' approach to helping patients change behavior. Am Fam Physician. 2000 Mar 1;61(5):1409-16. PMID 10735346
- [Background] Neighbors C, Dillard AJ, Lewis MA, Bergstrom RL, Neil TA. Normative misperceptions and temporal precedence of perceived norms and drinking. J Stud Alcohol. 2006 Mar;67(2):290-9. doi: 10.15288/jsa.2006.67.290. PMID 16562412
- [Background] Kahler CW, Hustad J, Barnett NP, Strong DR, Borsari B. Validation of the 30-day version of the Brief Young Adult Alcohol Consequences Questionnaire for use in longitudinal studies. J Stud Alcohol Drugs. 2008 Jul;69(4):611-5. doi: 10.15288/jsad.2008.69.611. PMID 18612578
- [Background] Moussas G, Dadouti G, Douzenis A, Poulis E, Tzelembis A, Bratis D, Christodoulou C, Lykouras L. The Alcohol Use Disorders Identification Test (AUDIT): reliability and validity of the Greek version. Ann Gen Psychiatry. 2009 May 14;8:11. doi: 10.1186/1744-859X-8-11. PMID 19442281
- [Background] Earleywine M, LaBrie JW, Pedersen ER. A brief Rutgers Alcohol Problem Index with less potential for bias. Addict Behav. 2008 Sep;33(9):1249-53. doi: 10.1016/j.addbeh.2008.05.006. Epub 2008 May 13. PMID 18547738
- [Background] Webb GR, Redman S, Gibberd RW, Sanson-Fisher RW. The reliability and stability of a quantity-frequency method and a diary method of measuring alcohol consumption. Drug Alcohol Depend. 1991 May;27(3):223-31. doi: 10.1016/0376-8716(91)90005-j. PMID 1884665
- [Background] Mange J, Mauduy M, Senemeaud C, Bagneux V, Cabe N, Jacquet D, Leconte P, Margas N, Mauny N, Ritz L, Gierski F, Beaunieux H. What really matters in binge drinking: A dominance analysis of binge drinking psychological determinants among University students. Addict Behav Rep. 2021 Apr 8;13:100346. doi: 10.1016/j.abrep.2021.100346. eCollection 2021 Jun. PMID 33997251
- [Background] Arterberry BJ, Martens MP, Cadigan JM, Smith AE. Assessing the Dependability of Drinking Motives via Generalizability Theory. Addict Res Theory. 2012 Oct 1;45(4):292-302. doi: 10.1177/0748175612449744. PMID 24696672
- [Background] Osberg TM, Atkins L, Buchholz L, Shirshova V, Swiantek A, Whitley J, Hartman S, Oquendo N. Development and validation of the College Life Alcohol Salience Scale: a measure of beliefs about the role of alcohol in college life. Psychol Addict Behav. 2010 Mar;24(1):1-12. doi: 10.1037/a0018197. PMID 20307107
- [Background] Xu S, Qiu D, Hahne J, Zhao M, Hu M. Psychometric properties of the short-form UCLA Loneliness Scale (ULS-8) among Chinese adolescents. Medicine (Baltimore). 2018 Sep;97(38):e12373. doi: 10.1097/MD.0000000000012373. PMID 30235699
- [Background] Zhong QY, Gelaye B, Zaslavsky AM, Fann JR, Rondon MB, Sanchez SE, Williams MA. Diagnostic Validity of the Generalized Anxiety Disorder - 7 (GAD-7) among Pregnant Women. PLoS One. 2015 Apr 27;10(4):e0125096. doi: 10.1371/journal.pone.0125096. eCollection 2015. PMID 25915929
- [Background] Carey KB, Carey MP, Maisto SA, Henson JM. Temporal stability of the timeline followback interview for alcohol and drug use with psychiatric outpatients. J Stud Alcohol. 2004 Nov;65(6):774-81. doi: 10.15288/jsa.2004.65.774. PMID 15700516
- See also: National Health and Nutrition Examination Survey Questionnaire — https://wwwn.cdc.gov/Nchs/Nhanes/Search/DataPage.aspx?Component=Dietary&Cycle=2009-2010.